CLINICAL TRIAL: NCT00018707
Title: Follow-up of Psychological and Neurocognitive Gulf War Outcome: Relation to Stress
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: MHBS-033-98F
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Gulf War Syndrome
MeSH Terms: conditions — Persian Gulf Syndrome

SUMMARY:
This is the follow-up to an observational epidemiological study of psychological and neuropsychological outcomes of deployed and non-deployed Gulf War-era veterans.

DETAILED DESCRIPTION:
Approximately 800 deployed and 250 nondeployed veterans were originally administered psychological assessment instruments shortly after the cessation of the Gulf War. These veterans are currently being followed to evaluate longer-term psychological outcomes in relation to war-zone stress, intervening life stress, and individual difference factors and personal resources, such as coping and social support.

Approximately 75 of these veterans, oversampled for post-traumatic stress disorder, were administered a specialized neuropsychological battery emphasizing attention and memory. This sample will also be followed to evaluate longitudinal neuropsychological outcome in relation to PTSD status.

A cross-sectional study will also be conducted examining visual, hierarchical attention in relation to PTSD diagnosis.

ELIGIBILITY:
Participation in Time 1 data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 1999-04; Study Completion 2003-03

CONTACTS AND LOCATIONS:
Locations (1):
- VA, New Orleans, New Orleans, Louisiana, United States